CLINICAL TRIAL: NCT05168202
Title: A Phase 1, Open-label, Dose Finding Study of CC-95251 Alone and in Combination With Antineoplastic Agents in Subjects With Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: A Study to Assess the Effect of CC-95251 in Participants With Acute Myeloid Leukemia and Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA059-001; 2021-002799-38 (EudraCT Number)
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia; AML; MDS; Hematologic Cancers; Leukemia; Anti-SIRPa antibody; CC-95251
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CC-95251 monotherapy (Experimental)
  Interventions: Drug: CC-95251
- CC-95251 + azacitidine (Experimental)
  Interventions: Drug: CC-95251; Drug: Azacitidine
- CC-95251 + azacitidine + venetoclax (Experimental)
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: CC-95251 — Specified dose on specified days
  Other Names: BMS-986351
  Arms: CC-95251 + azacitidine; CC-95251 monotherapy
Drug: Azacitidine — Specified dose on specified days
  Arms: CC-95251 + azacitidine
Drug: Venetoclax — Specified dose on specified days
  Arms: CC-95251 + azacitidine + venetoclax

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary clinical activity of CC-95251 alone and in combination with antineoplastic agents in participants with relapsed or refractory acute myeloid leukemia and relapsed or refractory and treatment-naive higher risk melodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

• Eastern Cooperative Oncology Group Performance Status of 0 to 2

For Parts A & B:

* Relapsed or refractory (R/R) acute myeloid leukemia (AML) as defined by the 2016 WHO Classification
* R/R myelodysplastic syndromes (MDS) as defined by the 2016 WHO Classification with intermediate, high or very high risk by Revised International Prognostic Scoring System (IPSS-R)

For Part C:

• Treatment-naïve (TN) (ie, previously untreated) MDS as defined by the 2016 WHO Classification with intermediate, high or very high risk by IPSS-R

For Part D:

• TN AML as defined by the 2016 WHO Classification, including secondary AML and therapy-related AML in participants who are ineligible (IE) for intensive chemotherapy (IC) and allogeneic hematopoietic stem cell transplant (HSCT)

Exclusion Criteria:

* Acute promyelocytic leukemia
* Immediately life-threatening, severe complications of leukemia such as disseminated/uncontrolled infection, uncontrolled bleeding, and/or uncontrolled disseminated intravascular coagulation
* Participants who have received prior treatment with a CD47 or SIRPα targeting agent
* Participant is on chronic systemic immunosuppressive therapy or corticosteroids
* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half-lives or 4 weeks prior to starting study treatment, whichever is shorter (relapsed or refractory participants only).
* Any condition including, active or uncontrolled infection, or the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study
* Pregnant or nursing participants.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (4):
  - Local Institution - 0030, Los Angeles, California
  - Local Institution - 0031, Palo Alto, California
  - Local Institution - 0047, Miami, Florida
  - Local Institution - 0001, Houston, Texas
- Australia (4):
  - Local Institution - 0027, Wollongong, New South Wales
  - Local Institution - 0006, Clayton, Victoria
  - Local Institution - 0005, Heidelberg, Victoria
  - Local Institution - 0037, Melbourne, Victoria
- Canada (4):
  - Local Institution - 0019, Edmonton, Alberta
  - Local Institution - 0011, Vancouver, British Columbia
  - Local Institution - 0010, Toronto, Ontario
  - Local Institution - 0038, Montreal, Quebec
- France (5):
  - Local Institution - 0040, Marseille
  - Local Institution - 0029, Nantes
  - Local Institution - 0020, Pessac
  - Local Institution - 0023, Toulouse
  - Local Institution - 0041, Villejuif
- Italy (3):
  - Local Institution - 0018, Meldola, Emilia-Romagna
  - Local Institution - 0026, Milan
  - Local Institution - 0017, Rozzano
- Norway (2):
  - Local Institution - 0025, Bergen
  - Local Institution - 0013, Oslo
- Spain (5):
  - Local Institution - 0032, Badalona, Barcelona [Barcelona]
  - Local Institution - 0039, Barcelona
  - Local Institution - 0036, Madrid
  - Local Institution - 0035, Salamanca
  - Local Institution - 0028, Santander
- Sweden (3):
  - Local Institution - 0021, Gothenburg
  - Local Institution - 0015, Lund
  - Local Institution - 0014, Stockholm
- United Kingdom (2):
  - Local Institution - 0044, Edinburgh, Midlothian
  - Local Institution - 0050, Oxford, Oxfordshire

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to a strategic re-evaluation and prioritization of the company's portfolio, this study was terminated early during dose escalation (Part A).
  No participants were enrolled in Parts B, C, and D because the study was terminated prior to the start of dose expansion.
Groups:
- Part A: Treatment 1: Monotherapy: CC-95251 20mg/kg
- Part A: Treatment 2: Monotherapy : CC-95251 30mg/kg
- Part A: Treatment 3: Combination : CC-95251 10mg/kg + Azacitidine 75 mg/m2
- Part A: Treatment 4: Combination : CC-95251 20mg/kg + Azacitidine 75 mg/m2
- Part A: Treatment 5: Combination : CC-95251 30mg/kg + Azacitidine 75 mg/m2
- Part A: Treatment 6: Triplet Combination : CC-95251 20mg/kg + Azacitidine 75 mg/m2 + Venetoclax
- Part A: Treatment 7: Triplet Combination : CC-95251 30mg/kg + Azacitidine 75 mg/m2 + Venetoclax
Period: Overall Study
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Started | 6 | 8 | 9 | 10 | 8 | 10 | 5
Completed (= Completed Study Treatment) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 9 | 10 | 8 | 10 | 5
Not completed — Progressive Disease | 4 | 4 | 2 | 3 | 2 | 3 | 2
Not completed — Adverse Event | 2 | 1 | 4 | 4 | 3 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1 | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Disease Relapse | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7 | Total
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (13.5) | 69.4 (10.82) | 68.3 (8.59) | 70.6 (4.25) | 67.5 (14.09) | 56.6 (16.53) | 65.4 (13.37) | 66.3 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 5 | 3 | 6 | 2 | 26
  Male | 2 | 6 | 5 | 5 | 5 | 4 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 3 | 5 | 6 | 4 | 3 | 6 | 4 | 31
  Unknown or Not Reported | 2 | 3 | 2 | 4 | 3 | 3 | 1 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 4 | 5 | 7 | 7 | 5 | 7 | 2 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 2 | 3 | 2 | 3 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DLTs
Description: A dose-limiting toxicity (DLT) is any treatment-related toxicity during Cycle 1 (Days 1-28, up to 42) not clearly due to illness or external causes. DLTs include:
  * Any Grade ≥3 non-hematologic toxicity, except specific reversible or manageable cases (e.g., IRR, nausea, diarrhea, fatigue, infection with leukemia, TLS, electrolyte imbalance, liver enzyme elevations, or rash).
  * Any confirmed Hy's law case (ALT/AST ≥3× ULN + bilirubin >2× ULN without cholestasis).
  * Hematologic toxicities: Grade 4 neutropenia/thrombocytopenia persisting at Day 28 without active AML/MDS; febrile neutropenia or Grade ≥3 thrombocytopenia with severe bleeding and prolonged myelosuppression (>42 days) without active leukemia.
  * Any adverse event requiring dose reduction in Cycle 1 unless clearly unrelated to the drug.
Time Frame: From Cycle 1 Day 1 to Cycle 1 Day 28 up to 42 post first dose of cycle 1 (upto 42 days)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Participants | 0 | 1 | 0 | 0 | 0 | 2 | 4

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.
Time Frame: From signing informed consent to 56 days post last dose (Approximately 30 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Participants | 6 | 8 | 8 | 9 | 8 | 10 | 5

3. Primary Outcome: Number of Participants With With Grade 3 or Higher Laboratory Abnormalities
Description: Clinical laboratory values from laboratories will be graded according to CTCAE Version 5 for applicable tests programmatically. For laboratory values that fall outside of the grade criteria of CTCAE Version 5, a Grade of 0 will be assigned. In addition, normal ranges will be used to determine the categories of High, Low, and Normal for laboratory tests that have no severity grade.
Time Frame: From signing informed consent to 56 days post last dose (Approximately 30 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Participants
  hemoglobin | 4 | 6 | 7 | 8 | 7 | 10 | 5
  platelet count | 5 | 8 | 9 | 10 | 8 | 10 | 5
  leukocytes | 5 | 5 | 6 | 9 | 7 | 9 | 4
  lymphocytes | 4 | 5 | 4 | 7 | 7 | 9 | 2
  neutrophils | 3 | 6 | 8 | 8 | 8 | 8 | 4
  Alanine aminotransferase | 0 | 1 | 1 | 0 | 0 | 3 | 1
  alkaline phosphatase | 0 | 1 | 0 | 0 | 0 | 0 | 1
  asparatate aminotransferase | 0 | 1 | 0 | 0 | 0 | 1 | 1
  bilirubin, total | 0 | 0 | 1 | 0 | 0 | 0 | 1
  creatinine | 0 | 0 | 0 | 1 | 0 | 0 | 0
  albumin | 0 | 0 | 1 | 1 | 0 | 1 | 0
  calcium, total | 0 | 0 | 0 | 1 | 0 | 0 | 0
  hyperkalemia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  hypocalcemia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  hypokalemia | 0 | 2 | 0 | 1 | 0 | 1 | 1
  hyponatremia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  potassium | 0 | 2 | 0 | 2 | 0 | 1 | 1
  sodium | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant ECG Abnormalities Presented as Adverse Events
Description: A single ECG will be performed in Screening, Cycle 1 Day 1 and 15, and Day 1 of Cycles ≥ 2. Investigators will make immediate clinical decisions based on their interpretation of the ECG results and provide their overall assessment.
Time Frame: From screening to 56 days post last dose (Approximately 29 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Participants
  Sinus Tachycardia | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Tachycardia | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Atrial Fibrillation | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Sinus Bradycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of ECOG Evaluations With Shift of ECOG Score of 3 or Greater.
Description: ECOG Scale was used to assess performance status. Grades: 0: Fully active, able to carry on all pre-disease performance without estriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead. Baseline value was defined as the last non-missing value on or before the day that first dose of study drug is administered; if multiple values are present for the same date, the average of these values will be used as the baseline.
Time Frame: From screening to 56 days post last dose (Approximately 29 months)
Population: Safety Population - Multiple ECOG evaluations were done throughout the study at different timepoints
Measure: Number; unit: ECOG Evaluations
Units Other Than Participants: ECOG Evaluation
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Number analyzed (ECOG Evaluation) | 27 | 41 | 29 | 45 | 45 | 29 | 15
ECOG Evaluations | 3 | 1 | 0 | 1 | 0 | 1 | 1

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Presented as AEs
Description: Vital sign measurements include: Weight (kg), Temperature (°C), Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Pulse (beats/min), Respiration Rate (breaths/min).
Time Frame: From signing informed consent to 56 days post last dose (Approximately 30 months)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 8 | 10 | 5
Participants
  Pyrexia | 0 | 1 | 1 | 2 | 3 | 4 | 1
  hypothermia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  hypertension | 0 | 0 | 1 | 0 | 1 | 2 | 0
  hypotension | 0 | 1 | 3 | 0 | 2 | 0 | 0
  weight decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0

7. Secondary Outcome: Cmax
Description: Maximum plasma concentration of drug
Time Frame: On Cycle 1 Day 1, C1D22 and C2D22.
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 10 | 5
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 8 | 5
  Cycle 1 Day 1 | 371.59 (25.14) | 510.58 (33.39) | 209.40 (14.13) | 428.72 (22.78) | 636.93 (7.80) | 418.39 (42.61) | 653.88 (10.36)
  Cycle 1 Day 22: number analyzed (Participants) | 4 | 7 | 6 | 8 | 7 | 7 | 3
  Cycle 1 Day 22 | 514.05 (25.01) | 773.08 (30.58) | 314.49 (16.76) | 641.78 (21.60) | 1055.99 (18.62) | 592.41 (50.25) | 1036.14 (28.08)
  Cycle 2 Day 22: number analyzed (Participants) | 3 | 4 | 6 | 6 | 5 | 4 | 1
  Cycle 2 Day 22 | 568.25 (32.29) | 1217.78 (19.11) | 318.09 (21.12) | 637.76 (21.01) | 1468.00 (18.85) | 833.06 (38.61) | 1470.00 (NA) — GCV not calculable due to only 1 participant analyzed

8. Secondary Outcome: Tmax
Description: Time to maximum plasma concentration (Tmax)
Time Frame: On Cycle 1 Day 1, C1D22 and C2D22.
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 10 | 5
hours
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 8 | 5
  Cycle 1 Day 1 | 2.33 [1.6 to 3.9] | 4.87 [2.1 to 7.2] | 1.80 [1.6 to 5.6] | 4.02 [2.5 to 6.0] | 5.47 [3.2 to 8.3] | 4.61 [2.1 to 22.3] | 4.78 [3.5 to 5.8]
  Cycle 1 Day 22: number analyzed (Participants) | 4 | 7 | 6 | 8 | 7 | 7 | 3
  Cycle 1 Day 22 | 1.93 [1.5 to 2.1] | 6.80 [2.1 to 7.6] | 3.17 [1.2 to 3.6] | 3.87 [2.0 to 22.6] | 5.88 [2.5 to 23.8] | 3.42 [1.6 to 23.9] | 6.75 [3.0 to 26.1]
  Cycle 2 Day 22: number analyzed (Participants) | 3 | 4 | 6 | 6 | 5 | 4 | 1
  Cycle 2 Day 22 | 3.78 [2.2 to 4.0] | 5.02 [2.3 to 7.1] | 3.51 [1.5 to 5.3] | 12.27 [1.9 to 69.6] | 3.28 [2.8 to 5.7] | 2.14 [1.8 to 3.8] | 3.37 [3.37 to 3.37]

9. Secondary Outcome: AUC(0-T)
Description: Area under the plasma concentration time-curve up to the last measurable concentration (AUC0-t)
Time Frame: On Cycle 1 Day 1, C1D22 and C2D22.
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 10 | 5
h*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 8 | 5
  Cycle 1 Day 1 | 27915.38 (25.74) | 37242.17 (41.18) | 13125.85 (48.00) | 23850.09 (50.97) | 49377.47 (10.90) | 28557.98 (61.21) | 42273.81 (28.09)
  Cycle 1 Day 22: number analyzed (Participants) | 4 | 7 | 6 | 8 | 7 | 7 | 3
  Cycle 1 Day 22 | 25766.21 (366.57) | 53952.86 (105.79) | 38363.45 (34.52) | 46250.05 (55.29) | 84673.85 (80.82) | 63857.81 (83.67) | 186843.83 (120.44)
  Cycle 2 Day 22: number analyzed (Participants) | 3 | 4 | 6 | 6 | 5 | 4 | 1
  Cycle 2 Day 22 | 42891.42 (38.09) | 54797.36 (205.65) | 37672.97 (30.69) | 54425.19 (131.05) | 116229.58 (23.27) | 74865.57 (104.46) | 137581.5 (NA) — GCV not calculable due to only 1 participant analyzed

10. Secondary Outcome: AUC(TAU)
Description: Area under the plasma concentration time-curve during a dosing interval (AUCtau)
Time Frame: On Cycle 1 Day 1, C1D22 and C2D22.
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 10 | 5
h*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 6 | 7 | 8 | 8 | 7 | 4
  Cycle 1 Day 1 | 27915.38 (25.74) | 39145.67 (33.39) | 15987.61 (16.16) | 28817.51 (27.62) | 49377.47 (10.90) | 29931.17 (64.80) | 46778.93 (18.30)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 4 | 6 | 5 | 5 | 7 | 3
  Cycle 1 Day 22 | 48306.42 (48.94) | 87419.67 (68.23) | 34295.76 (16.51) | 64776.31 (16.33) | 120818.65 (32.18) | 57119.56 (67.28) | 109428.93 (41.91)
  Cycle 2 Day 22: number analyzed (Participants) | 2 | 2 | 6 | 3 | 4 | 3 | 1
  Cycle 2 Day 22 | 48436.92 (44.72) | 128864.45 (8.24) | 37672.97 (30.69) | 89459.57 (19.99) | 119737.08 (25.79) | 114221.87 (19.11) | 137581.85 (NA) — GCV not calculable due to only 1 participant analyzed

11. Secondary Outcome: Cmin
Description: Minimum serum concentration
Time Frame: On Cycle 1 Day 1, C1D22 and C2D22.
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
Number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 10 | 5
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 7 | 9 | 10 | 8 | 8 | 5
  Cycle 1 Day 1 | NA (NA) — Below the limit of quantification | 1.96 (NA) — Below the limit of quantification | NA (NA) — Below the limit of quantification | 140.00 (NA) — Below the limit of quantification | NA (NA) — Below the limit of quantification | NA (NA) — Below the limit of quantification | 0.47 (NA) — Below the limit of quantification
  Cycle 1 Day 22: number analyzed (Participants) | 4 | 7 | 6 | 8 | 7 | 7 | 3
  Cycle 1 Day 22 | 149.97 (50.58) | 213.59 (104.90) | 109.90 (40.52) | 153.17 (97.33) | 342.42 (39.35) | 167.12 (89.50) | 336.79 (54.07)
  Cycle 2 Day 22: number analyzed (Participants) | 3 | 4 | 6 | 6 | 5 | 4 | 1
  Cycle 2 Day 22 | 171.28 (48.96) | 588.04 (36.19) | 135.10 (44.61) | 225.45 (37.09) | 573.75 (46.78) | 291.15 (94.88) | 545.00 (NA) — Below the limit of quantification

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events and All Cause Mortality: (Approximately 30 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Part A: Treatment 1: Monotherapy : CC-95251 20mg/kg
Arm/Group | Part A: Treatment 1 | Part A: Treatment 2 | Part A: Treatment 3 | Part A: Treatment 4 | Part A: Treatment 5 | Part A: Treatment 6 | Part A: Treatment 7
All-Cause Mortality (participants affected / at risk) | 6/6 | 7/8 | 6/9 | 9/10 | 6/8 | 8/10 | 3/5
Serious Adverse Events (participants affected / at risk) | 6/6 | 7/8 | 8/9 | 7/10 | 7/8 | 10/10 | 5/5
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 7/9 | 9/10 | 7/8 | 10/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment 1 (N=6) | Part A: Treatment 2 (N=8) | Part A: Treatment 3 (N=9) | Part A: Treatment 4 (N=10) | Part A: Treatment 5 (N=8) | Part A: Treatment 6 (N=10) | Part A: Treatment 7 (N=5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 5 | 3 | 1 | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 2
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 3 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningorrhagia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment 1 (N=6) | Part A: Treatment 2 (N=8) | Part A: Treatment 3 (N=9) | Part A: Treatment 4 (N=10) | Part A: Treatment 5 (N=8) | Part A: Treatment 6 (N=10) | Part A: Treatment 7 (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 3 | 3 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 3 | 1 | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 5 | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 4 | 2 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3 | 5 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosa haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 2 | 2 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 3 | 1 | 0 | 4 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 1
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Medical device site thrombosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 3 | 3 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cystitis escherichia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vascular access site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1 | 2 | 1 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0 | 0 | 1 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1 | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 2 | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 2 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to a strategic re-evaluation and prioritization of the company's portfolio, this study was terminated early during dose escalation (Part A) and prior to the start of dose expansion (Parts B, C, and D) with no relation to any safety issues associated with the use of CC-95251. Due to this termination, secondary efficacy endpoints, which were for these dose expansion cohorts, were not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT05168202/Prot_SAP_000.pdf